CLINICAL TRIAL: NCT04367714
Title: Antistof Respons Mod SARS-CoV-2 Hos Dialysepatienter i Forbindelse Med COVID-19
Brief Title: Antibody Response Against SARS-CoV-2 in Dialysis Patients During COVID-19
Acronym: COVCKD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region MidtJylland Denmark (Other)
Collaborators: Aarhus University Hospital (Other); Central Jutland Regional Hospital (Other); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Frank Mose, MD PhD, Region MidtJylland Denmark
Other Study IDs: FHM-1-2020
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: COVID; Terminal Renal Insufficiency
Keywords: COVID-19; CKD 5
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples With DNA — Samples for determination of antibodies, cytokines, RNA and DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Determination of IgM and IgG antibodies against SARS-CoV-2 in dialysis patients by continous monitoring in the period from March 2020 to december 2020

DETAILED DESCRIPTION:
Blood samples are collected every 14 days

ELIGIBILITY:
Inclusion Criteria:

* Dialysis

Exclusion Criteria:

* Not willing to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dilaysis patients on 3 Danish center in Jutland
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-03-15 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
AAntibody response | 1 year
  IgM and IgG against SARS-CoV-2

CONTACTS AND LOCATIONS:
Locations (1):
- Godstrup Hospital, Herning, Denmark

IPD SHARING:
Plan to Share IPD: No